CLINICAL TRIAL: NCT01501461
Title: An Open-label, Non-Randomized, Multi-Center Study to Assess the Safety and Effects of Intra-venous Implantation of Autologous Adipose-Derived Stem Cells in Patients With Frailty Syndrome
Brief Title: Study to Assess the Safety and Effects of Autologous Adipose-Derived Stem Cells in Patients With Frailty Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Company dissolved
Sponsor: Ageless Regenerative Institute (Industry)
Collaborators: Instituto de Medicina Regenerativa (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADI-ME-FS-001
Record Dates: First submitted 2011-10-03; First posted 2011-12-29 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2017-11

CONDITIONS: Frailty Syndrome
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Harvesting and implantation of stem cells — The adipose tissue specimen will be collected from the patient's abdomen or applicable area using tumescent syringe liposuction. The adipose tissue is transferred to the laboratory for separation of the adipose tissue-derived stem cells, which are then transferred for injection intravenously.

SUMMARY:
The intent of this clinical study is to answer the questions:

1. Is the proposed treatment safe
2. Is treatment effective in improving the health of patients with human frailty syndrome.

DETAILED DESCRIPTION:
This will be an open-label, non-randomized multi-center patient sponsored study of Autologous Adipose-Derived Stem Cells (ASC) implantation after liposuction using an IV delivery system. ASCs will be derived from the patient's adipose-derived tissue. Liposuction using local anesthesia and syringe collection will be performed to collect the adipose tissue specimen for subsequent processing to isolate the stem cells. The cells will be delivered intravenously.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females Age >55.
* Frailty syndrome defined by:

BMD< T-1 (Based on QCT results) Body Mass: males <8% or >17% fat, females<10% or>24% fat (Lean Body Mass=Total Body Mass- %Body Fat)

* Ability to participate in the short physical performance battery
* Up to date on all age and gender appropriate cancer screening per American Cancer Society

Exclusion Criteria:

* Life expectancy < 6 months due to concomitant illnesses.
* Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
* Active infectious disease patients known to have tested positive for HIV, HTLV, HBV, HCV, CMV (IgM > IgG) and/or syphilis. will have an expert consulted as to patient eligibility based on the patient's infectious status
* Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
* Patients on chronic immunosuppressive transplant therapy
* Active clinical infection being treated by antibiotics within one week of enrollment.
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* History of cancer (other than non-melanoma skin cancer or in-situ cervical cancer) in the last five years.
* Unwilling and/or not able to give written informed consent.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05-01; Primary Completion 2017-05-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Improvement in Physical Performance Test (PPT) Results | 3 months
Number of Adverse Events Reported | up to 6 months
  The safety of adipose-derived stem cell injection will be evaluated by assessment of the frequency and nature of adverse events occurring during the study injection and up to the 6-month period following treatment.
Improvement in Physical Performance Test (PPT) Results | 6 months
Improved body composition/bone density compared to baseline | 3 months
Improved body composition/bone density compared to baseline | 6 months
Quality of life is improved compared to baseline | 3 months
Quality of life is improved compared to baseline | 6 months

SECONDARY OUTCOMES:
Improved exercise capacity compared to baseline | 3 months
Improved exercise capacity compared to baseline | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clemente Zuniga, MD, Principal Investigator — Instituto de Medicina Regenerativa; Jesus A Perez, MD, Principal Investigator — Instituto de Medicina Regenerativa
Locations (1):
- Instituto de Medicina Regenerativa, Tijuana, Estado de Baja California, Mexico